CLINICAL TRIAL: NCT02739789
Title: Activating and Identifying Neural Responses to Social Rejection: a Combined Transcranial Direct Current Stimulation (tDCS) and Functional Magnetic Resonance Imaging (fMRI) Study
Brief Title: Activating and Identifying Neural Responses to Social Rejection: a Combined tDCS and fMRI Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, David Hsu, Assistant Professor of Psychiatry, Stony Brook University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: SBU Psychiatry Pilot
Record Dates: First submitted 2016-04-01; First posted 2016-04-15 (Estimated); Results first posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-06

CONDITIONS: Healthy
Keywords: tDCS rejection affect mood fMRI
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: within-subjects crossover design
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham tDCS (Sham Comparator): tDCS stimulation will be administered over the brain area of interest, but will be shorter in duration than the "active" treatment
  Interventions: Device: Sham tDCS
- Active tDCS (Active Comparator): tDCS stimulation will be administered over the brain area of interest
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — tDCS
  Arms: Active tDCS
Device: Sham tDCS — Sham tDCS
  Arms: Sham tDCS

SUMMARY:
This research study identifies neural pathways regulating negative moods during rejection by combining transcranial direct current stimulation (tDCS) and fMRI in a sample of healthy controls.

DETAILED DESCRIPTION:
Aim 1: To test the behavioral effects of tDCS during social rejection. The first step will be to obtain behavioral effects of transcranial direct current stimulation (tDCS) during social rejection without functional magnetic resonance imaging (fMRI). Whereas previous studies used "Cyberball" (a computerized ball-tossing game that simulates social exclusion), we will use the Social Feedback Task. This task was created by Dr. Hsu to be more ethologically-relevant, has been shown to sustain negative moods during rejection and activates the right ventral lateral prefrontal cortex (rVLPFC) (preliminary fMRI data from 50 healthy controls in Dr. Hsu's previous study). Anodal tDCS will be applied over the right or left VLPFC to measure changes in mood during rejection and neutral conditions. Depending on results, alternate regions in separate subjects may also be stimulated: dorsolateral prefrontal cortex, insula, anterior cingulate cortex, pre-supplementary, and supplementary motor area [all regions may be right or left hemisphere]. All of these regions have been shown to be involved in emotion regulation. Questionnaires will be given before, during, and after the task to assess cognitive and emotional states.

Aim 2: To identify neural pathways regulating negative moods during social rejection, using tDCS for activation and fMRI for assessment. Using a cross-over, sham-controlled design similar to previous tDCS+fMRI studies, we will measure the effects of anodal tDCS over the right or left VLPFC on neural activity and negative mood during rejection and neutral conditions. Alternate regions in separate subjects may also be stimulated including the dorsolateral prefrontal cortex, insula, anterior cingulate cortex, pre-supplementary, and supplementary motor area [all regions may be right or left hemisphere]. All of these regions have been shown to be involved in emotion regulation.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or females between 18 and 25 years old
2. No diagnosis on Axis I by Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders IV. No current, or within the past 5 years.
3. Not currently in a romantic relationship
4. Ability to understand and follow instructions and oriented to name, time, and place.
5. No additional neurologic or psychiatric disorders
6. No current use of psychotropic drugs or during past 3 months (except marijuana and alcohol)
7. No current use of marijuana or during past 3 weeks
8. Not currently abusing alcohol
9. No history of alcohol or drug dependence within past 5 years
10. A negative urine pregnancy and toxicology screen. Verbal affirmation will be obtained (i.e., "not pregnant" and "not currently using psychotropic drugs or during the past 3 months") during the Screening Visit (Day 1). Urine screen will be obtained on Days 2 and 3. If subject reports that there is a "possibility that she is pregnant" on Day 1 (Screening Visit) a urine pregnancy screen will be performed on that day.
11. (Women): If stopped or started oral contraceptives recently, at least 60 days on/off oral contraceptives.

Exclusion Criteria:

1. Left-handed or ambidextrous
2. Metallic dental implants
3. Metallic objects in the brain/skull
4. Medical device implants
5. Implanted electronic devices
6. History of seizures
7. History of strokes
8. Unexplained loss of consciousness
9. Frequent or severe headaches or neck pain
10. Clinically significant, uncontrolled liver, kidney, cardiac, or pulmonary disease
11. Terminal medical diagnosis consistent with survival < 1 year
12. Pregnancy; childbirth or miscarriage within 6 months, breastfeeding within 6 months of recruitment
13. Serious mental impairment. Mini mental state exam of < 23/30
14. Chronic skin disease
15. Previous experience with transcranial direct current stimulation (tDCS)
16. Regular tobacco use or tobacco use within past month
17. If using hormonal birth control, taking progestin-only pills (e.g., Cerazette, Ovrette), or Intrauterine devices (Mirena, Skyla), since progestin-only birth controls are more likely to cause mood swings.

Addition Exclusion Criteria for participating in fMRI:

1. Metal anywhere in the body
2. Weight over 250 pounds, or girth size incompatible for scanner bore.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2018-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David T Hsu, PhD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a within-subjects design, thus every subject received both active and sham conditions
Groups:
- Sham tDCS First, Then Active tDCS: Sham transcranial direct current stimulation (tDCS) on first scan day: tDCS stimulation will be administered over the brain area of interest, but will be shorter in duration than the "active" treatment.
  Active tDCS on second scan day: tDCS stimulation will be administered over the brain area of interest.
- Active tDCS First, Then Sham tDCS: Active tDCS on first scan day: tDCS stimulation will be administered over the brain area of interest.
  Sham tDCS on second scan day: tDCS stimulation will be administered over the brain area of interest, but will be shorter in duration than the "active" treatment.
Period: First fMRI Scan
Arm/Group | Sham tDCS First, Then Active tDCS | Active tDCS First, Then Sham tDCS
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0
Period: ~1 Week Waiting Period
Arm/Group | Sham tDCS First, Then Active tDCS | Active tDCS First, Then Sham tDCS
Started | 9 | 10
Completed | 9 | 7
Not Completed | 0 | 3
Period: Second fMRI Scan
Arm/Group | Sham tDCS First, Then Active tDCS | Active tDCS First, Then Sham tDCS
Started | 9 | 7
Completed | 9 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham tDCS | Active tDCS | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.89 (2.37) | 21.71 (1.80) | 21.81 (2.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 5 | 3 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White or Caucasian | 5 | 3 | 8
  Race/Ethnicity: Black or African American | 0 | 1 | 1
  Race/Ethnicity: Hispanic or Latino | 0 | 0 | 0
  Race/Ethnicity: Asian | 3 | 3 | 6
  Race/Ethnicity: American Indian or Alaskan Native | 0 | 0 | 0
  Race/Ethnicity: Other or mixed | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Blood Oxygen Level Dependent (BOLD) Signal Changes (in Arbitrary Units)
Description: Images from fMRI scans for each participant are preprocessed (e.g., realigned, normalized, smoothed). Changes in BOLD signal are modeled for rejection and acceptance vs neutral blocks, and contrast images are created. These contrast images are used to compare tDCS vs sham for each subject in a within-subjects analysis. BOLD responses are reported as arbitrary units (i.e., change from sham stimulation). Regions of interest include left and right ventrolateral prefrontal cortex (VLPFC), left and right nucleus accumbens (NAcc), left and right amygdala (Amyg), left and right anterior insula (AI), left and right dorsal anterior cingulate cortex (dACC).
Time Frame: 1-3 weeks
Measure: Mean (Standard Deviation); unit: Arbitrary units
Arm/Group | Sham tDCS | Active tDCS
Number analyzed (Participants) | 16 | 16
Arbitrary units
  left VLPFC (Rejection-Neutral) | .57 (.77) | .66 (.80)
  right VLPFC (Rejection-Neutral) | .25 (.49) | .29 (.38)
  left VLPFC (Acceptance-Neutral) | .67 (.84) | .33 (.77)
  right VLPFC (Acceptance-Neutral) | .40 (1.14) | .31 (.72)
  left NAcc (R-N) | .01 (.25) | .18 (.42)
  right NAcc (R-N) | .05 (.30) | .24 (.53)
  left NAcc (A-N) | .09 (.38) | .27 (.38)
  right NAcc (A-N) | .17 (.38) | .34 (.58)
  left Amyg (R-N) | .2 (.36) | .39 (.45)
  right Amyg (R-N) | .19 (.41) | .35 (.52)
  left Amyg (A-N) | .12 (.43) | .11 (.23)
  right Amyg (A-N) | .07 (.43) | .19 (.38)
  left AI (R-N) | .32 (.49) | .38 (.53)
  right AI (R-N) | .28 (.49) | .23 (.61)
  left AI (A-N) | .36 (.60) | .32 (.44)
  right AI (A-N) | .21 (.86) | .17 (.41)
  left dACC (R-N) | .04 (.60) | .25 (.67)
  right dACC (R-N) | .13 (.45) | .21 (.72)
  left dACC (A-N) | .09 (.6) | .42 (.62)
  right dACC (A-N) | .06 (.59) | .32 (.67)

2. Primary Outcome: Change in Positive and Negative Affect Scale (During fMRI)
Description: Change in emotion will be measured on the "Positive and Negative Affect Scale." During Rejection, Acceptance, and Neutral conditions, participants rate how much they feel "sad," "rejected," "happy," and "accepted" on a visual analog scale from "not at all" (minimum score of "0") to "extremely" (maximum score of "100").
  Scores for "sad" were averaged with "rejected," and scores for "happy" were averaged with "accepted." The averaged scores during Neutral were subtracted from Rejection and Acceptance to derive the outcome measures.
  Higher outcome measure score means that the participant felt more of that particular emotion during a particular condition (minus neutral). Thus, a higher score for "happy and accepted" during the Acceptance-Neutral condition means a better outcome. Similarly, a lower score for "happy and accepted' during Rejection-Neutral condition means a worse outcome.
Time Frame: 1-3 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham tDCS | Active tDCS
Number analyzed (Participants) | 16 | 16
score on a scale
  Rejection-Neutral conditions (sad and rejected) | 14.06 (18.82) | 12.81 (14.72)
  Acceptance-Neutral conditions (sad and rejected) | 6.00 (20.63) | -3.33 (13.84)
  Rejection-Neutral conditions (happy and accepted) | -10.94 (22.89) | -5.31 (20.37)
  Acceptance-Neutral conditions (happy and accepted) | 0 (22.20) | 12.00 (25.48)

3. Primary Outcome: Change in the Single-item Self-Esteem Scale (During fMRI)
Description: Change in self-esteem will be measured on the "Single-item Self-Esteem Scale." During Rejection, Acceptance, and Neutral conditions, participants respond to the item "I have high self-esteem" on a visual analog scale from "not at all true of me" (minimum score of "0") to "very true of me" (maximum score of "100").
  Scores during Neutral were subtracted from Rejection and Acceptance to derive the outcome measures.
  Higher outcome measure score means that the participant had more self-esteem, and thus a better outcome, during a particular condition (minus neutral).
Time Frame: 1-3 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham tDCS | Active tDCS
Number analyzed (Participants) | 16 | 16
score on a scale
  Rejection-Neutral conditions | -5.33 (18.46) | -2.67 (21.54)
  Acceptance-Neutral conditions | 0.71 (12.69) | 8.57 (28.78)

4. Primary Outcome: Change in Desire for Social Interaction Scale (During fMRI)
Description: Change in Desire for Social Interaction will be measured on the "Desire for Social Interaction Scale." During Rejection, Acceptance, and Neutral conditions, participants respond to four items measuring desire for social interaction (e.g., "I would enjoy social interaction right now") on a visual analog scale from "very slightly or not at all" (minimum score of "0") to "extremely" (maximum score of "100").
  Scores during Neutral were subtracted from Rejection and Acceptance to derive the outcome measures.
  Higher outcome measure score means that the participant had greater desire for social interaction, and thus a better outcome, during a particular condition (minus neutral).
Time Frame: 1-3 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sham tDCS | Active tDCS
Number analyzed (Participants) | 16 | 16
score on a scale
  Rejection-Neutral conditions | -16.88 (35.72) | -13.75 (30.30)
  Acceptance-Neutral conditions | -2.00 (14.24) | 1.33 (19.22)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the duration of time over which each participant was assessed. This was an average of 30 days (standard deviation = 16 days, range = 14 - 74 days).
Groups:
- Sham tDCS: Sham tDCS: tDCS stimulation will be administered over the brain area of interest, but will be shorter in duration than the "active" treatment.
  All participants received sham tDCS, either on the first or second scan day.
- Active tDCS: Active tDCS: tDCS stimulation will be administered over the brain area of interest.
  All participants received active tDCS, either on the first or second scan day.
Arm/Group | Sham tDCS | Active tDCS
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/89/NCT02739789/Prot_SAP_ICF_000.pdf